CLINICAL TRIAL: NCT00915746
Title: An Open-Label Drug-Drug Interaction Study to Assess the Effect of Ketoconazole on the Pharmacokinetics of JNJ-31001074 in Healthy Subjects
Brief Title: A Drug Interaction Study of JNJ-31001074 and Ketoconazole in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Clinical Leader, Psychiatry, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CR016342
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Last update posted 2010-04-30 (Estimated); Status verified 2010-04

CONDITIONS: Healthy; Pharmacokinetics; Drug Interactions
Keywords: Phase I; ketoconazole; CYP3A4 inhibitor; drug interaction; metabolism; Healthly Volunteer; JNJ-31001074
MeSH Terms: interventions — bavisant; Ketoconazole

INTERVENTIONS:
Drug: JNJ-31001074; ketoconazole

SUMMARY:
This is an open-label (both the physician and healthy volunteer know which treatment will be administered) study to assess the pharmacokinetics (process by which JNJ-31001074 is absorbed, distributed, metabolized, and eliminated by the body) of JNJ-31001074 when taken alone and in combination with ketoconazole. The study consists of three phases: a screening phase to determine eligibility, an open-label treatment phase consisting of three periods and an end-of study/early withdrawal assessment phase.

DETAILED DESCRIPTION:
This is an open-label (both the physician and healthy volunteer know which treatment will be administered), sequential design (one after the other) study to assess the pharmacokinetics (process by which JNJ-31001074 is absorbed, distributed, metabolized, and eliminated by the body) of JNJ-31001074 when taken alone and in combination with ketoconazole. The study consists of three phases: a screening phase to determine eligibility, an open-label treatment phase consisting of three periods and an end-of-study/early withdrawal assessment phase. During the screening phase, healthy volunteers will be evaluated to see if they meet selection criteria as specified in the protocol. Healthy volunteers who meet these criteria will report to the study center on Day -1. Volunteers will be admitted to the study center and will fast (no food or beverages) overnight for at least 10 hours. Volunteers will remain at the study center for 11 days. The open-label treatment phase consists of three periods. In Period 1, a single-dose of JNJ-31001074 10 mg will be administered on Day 1, followed by three days of multiple blood sampling (Days 1-3). In Period 2 (Days 4-6), 400 mg ketoconazole will be administered on each day just prior to which predose blood samples are taken. In Period 3 (Days 7-11), JNJ-31001074 10 mg and ketoconazole 400 mg will be administered together on Day 7, followed by four days of multiple blood sampling. Ketoconazole will also be administered on Day 8 and Day 9 of Period 3. No study drug will be administered on Days 2 and 3 of Period 1, and Days 10 and 11 of Period 3. The end-of-study phase assessments will be performed after the completion of the four day blood sampling on Day 11. Safety and tolerability will be assessed throughout the volunteer's participation. Volunteers will be instructed to report any adverse events that occur up to 30 days after their last dose of study drug. The maximum study duration for each volunteer is expected to be 32 days. JNJ-31001074 10 mg will be administered orally on Days 1 and 7; ketoconazole 400 mg will be administered orally on Days 4, 5, 6, 7, 8, and 9.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer between the ages of 18-55
* if a woman, must be of non childbearing potential (ie, post menopausal or surgically sterile) and have a negative pregnancy test
* body mass index between 18-30
* body weight greater than or equal to 50 kilograms
* blood pressure between 90 and 140 mgHg systolic and no higher than 90 mgHg diastolic
* nonsmoker

Exclusion Criteria:

* History of or current clinically significant medical illness
* clinically significant abnormal laboratory value(s)
* clinically significant abnormal physical examination, vital signs or electrocardiogram
* pregnant, lactating or completed last term pregnancy within six months of screening
* use of any prescription or non prescription medication except for paracetamol (acetaminophen/TYLENOL), bisphosphonates (drugs to treat osteoporosis), hormone replacement therapy within 14 days of first dose of study medication
* history of drug or alcohol abuse
* history of smoking or use of nicotine-containing substances within the previous two months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-11; Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The primary objective is to assess the effects of repeated daily administration of 400 mg of ketoconazole on the single-dose pharmacokinetics of JNJ-31001074 in healthy volunteers | Multiple blood samples will be obtained over the 11 day open-label treatment phase

SECONDARY OUTCOMES:
To assess the safety and tolerability of JNJ-31001074 with and without coadministration of ketoconazole | up to 32 days (including a 21 day screening phase)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.